CLINICAL TRIAL: NCT02345876
Title: Asymmetry, Auditory Processing and Reading Skills in Phonological Dyslexic Children Compared to Average-reading Children
Brief Title: Maturation of Auditory Processing in Children With Dyslexia Compared to Average-reading Children
Acronym: ASTRAUCOLE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-799
Record Dates: First submitted 2014-12-09; First posted 2015-01-26 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Dyslexia
Keywords: Dyslexia, Medial olivocochlear system, Maturation, Auditory Processing
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dyslexic children: Longitudinal follow-up without intervention
  Interventions: Other: no intervention
- Normal reading children: Longitudinal follow-up without intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The hypothesis of central auditory processing disorders has been advanced to explain the anomalies of the grapheme/phoneme combination in some dyslexia. These phonological disorders may be linked to abnormalities of the efferent (medial olivocochlear) system modulation and of cortical asymmetry. Indeed, the efferent system has an asymmetry in relation to handedness. Thus, in right-handed subject, it is predominant on the right side. In contrast, in the subject-handed dyslexic, the efferent system tends to be right-lateralized or non-lateralized. However, after an audio-visual training, normal lateralization can appear. This maturation of the efferent system lateralization during reading acquisition seems to have a particular profile in dyslexics with phonological disorder, especially if it is persistent. This finding allows to consider new prognostic evaluation and speech therapy rehabilitation in the dyslexic child.

ELIGIBILITY:
Common inclusion criteria

* Native French speaker and french education
* No medical treatment for behavior or neurological disorders (as epilepsy)
* Normal or corrected vision
* Right-handed children (Edinburgh tets (Oldfield, 1971): >+50%)
* Normal ORL examination
* No hearing loss : hearing thresholds not above 15 dB between 250 and 4 000 Hz
* Presence of Otoacoustic Emissions (Total amplitude < 5 dB or SNR > 3dB for at least 3 frequency bands between 1 and 4 kHz)
* Normal level of intellectual development
* Regular school attendance

For the normal reading children

* Aged from 6 to less than 11
* Normal reading level

For the dyslexic children

* Aged from 8 to less than 11
* Diagnostic of dyslexia made by a complet check-up during the 6 last months before the inclusion

Exclusion Criteria

* Neurological or psychiatric disease incompatible with the testing procedure
* Ear disease during more than 6 months
* Normal reading children who have repeat a year
* Previous speech therapy for normal reading children
* Not corrected visual acuteness
* Schooling in a foreign language
* Foreign language spoken at home with both parents
* Known hearing deficit
* Invalid social security

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: For the dyslexic children: primary care clinic and speech therapists For the normal reading children : elementary schools of Lyon and Clermond-Ferrand and their suburbs
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Change of The Asymmetry Index of the efferent system at 2 years interval | Day 1 and then at least 2 years (± 4 weeks)
  The change of the Asymmetry Index of the efferent system The Asymmetry Index is the difference between the equivalent attenuation measured on the right ear and the left ear. Evoked otoacoustic emissions were recorded monaurally at five stimulus intensities ranging from 57 to 69 dB SPL in 3 dB steps, in random presentation order, with and without contralateral acoustic stimulation consisting of 30 dBSPL continuous broadband noise (speech-like noise) produced by an audiometer

SECONDARY OUTCOMES:
Change in the level of reading skill | Day 1 and then at least 2 years (± 4 weeks)
  Behavioral measure
Change in the percentage of correct answers obtained during a speech perception test in silence and noise. | Day 1 and then at least 2 years (± 4 weeks)
  Oral repetition of VCV
Change in percentage of correctly repeated stimuli which have been heard in both ears (binaural integration with divided attention) or in one indicated ear (binaural separation with selective attention) | Day 1 and then at least 2 years (± 4 weeks)
  Presentation of different speech material to both ears simultaneously

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Hospitzlier Le Vinatier, Bron
  - Service ORL CHU Montpied, Clermont-Ferrand
  - Service d'Audiologie et Explorations Orofaciales Centre de Référence des Troubles des Apprentissages, Lyon